CLINICAL TRIAL: NCT00218543
Title: Atomoxetine Treatment for Cocaine Abuse and Adult Attention-Deficit Hyperactivity Disorder (ADHD): A Preliminary Open Trial
Brief Title: Atomoxetine for Treating Cocaine Abuse in Adults With Attention Deficit Hyperactivity Disorder (ADHD)
Acronym: Atom
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Frances R Levin, Director of Substance Use Disorder, New York State Psychiatric Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: #4611; P50DA009236 (NIH); P50-09236-12; DPMC
Record Dates: First submitted 2005-09-20; First posted 2005-09-22 (Estimated); Results first posted 2012-07-04 (Estimated); Last update posted 2019-04-24 (Actual); Status verified 2019-04

CONDITIONS: Attention Deficit Disorder With Hyperactivity; Cocaine-Related Disorders
Keywords: ADHD; Cocaine Abuse
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Cocaine-Related Disorders | interventions — Atomoxetine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Atomoxetine (Experimental): Atomoxetine
  Interventions: Drug: Atomoxetine

INTERVENTIONS:
Drug: Atomoxetine — At the start of week 7, patients will be maintained at 80 mg/day or increased to the maximal dose of 100 mg/day if less than a 50% reduction of symptoms on the ADHD Rating Scale occurs, and if the patient is tolerating the medication well.

SUMMARY:
Studies have shown that individuals with attention deficit hyperactivity disorder (ADHD) are at greater risk for having a substance use disorder compared to people who do not have ADHD. Rates of cocaine abuse in adults with ADHD are significantly higher than they are in adults who do not have ADHD. Some clinicians suggest that adults with ADHD may abuse cocaine in order to self-medicate their ADHD symptoms. Atomoxetine is a drug that has been effective in treating ADHD. This study will evaluate the effectiveness of atomoxetine in reducing cocaine use in people with ADHD who abuse cocaine.

DETAILED DESCRIPTION:
ADHD is a neurologic disorder that is thought to be caused by chemical imbalances of certain neurotransmitters in the brain. The disorder can cause inattention, hyperactivity, and impulsivity. Cocaine abuse rates in adults with ADHD are significantly higher than they are in adults who do not have the disorder. This may be reflective of an attempt by individuals with ADHD to self-treat symptoms. Atomoxetine is an FDA-approved drug that is used to increase the ability to pay attention and decrease impulsiveness and hyperactivity in children and adults with ADHD. The drug is in a class of medications called selective norepinephrine reuptake inhibitors and works by increasing the levels of norepinephrine, a natural substance in the brain that affects a person's attention and impulsivity. It is possible that reducing ADHD symptoms in cocaine abusers with ADHD will help decrease their need for cocaine. This study will evaluate the effectiveness of atomoxetine in reducing cocaine use in people with ADHD who abuse cocaine.

Participants in this open label study will receive atomoxetine for 12 weeks, and will take one dose each morning for the duration of the study. Doses will be increased gradually to minimize side effects and enhance treatment compliance. In addition, all participants will receive individualized relapse prevention therapy once weekly. Participants will be required to report to the study site three times a week to receive medication, complete questionnaires regarding ADHD symptoms and substance use behavior, and provide a urine sample while being supervised by study staff. Also, vital signs will be monitored and medication side effects will be assessed at each visit. Participants will report to the study site 6 months after starting in the study for a follow-up visit, at which time ADHD symptoms, substance use behavior, and social functioning will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Meets DSM-IV criteria for cocaine dependence and adult ADHD
* Describes cocaine as the primary drug of abuse
* Meets DSM-IV criteria for cocaine dependence

Exclusion Criteria:

* Meets DSM-IV criteria for current Axis I psychiatric disorders that require a psychiatric intervention (except ADHD or substance abuse)
* Current major depression
* Unstable physical disorders that might make participation unsafe (e.g., uncontrolled high blood pressure and tachycardia [systolic blood pressure greater than 150 mm Hg, diastolic blood pressure greater than 90 mm Hg, or a sitting heart rate greater than 100])
* Acute hepatitis (individuals with chronic mildly elevated transaminase levels of less than 2 or 3 times the normal limit are not excluded)
* Diabetes
* Coronary vascular disease, as indicated by a history or suspected by an abnormal electrocardiogram
* History of cardiac symptoms
* History of seizures
* Narrow angle glaucoma
* Use of monoamine oxidase inhibitors (MAOIs) within 2 weeks of starting treatment with atomoxetine
* Currently taking prescribed psychotropic medications
* Currently taking medications for the treatment of ADHD
* Known sensitivity to atomoxetine
* Current suicidal ideation or history of suicidal or homicidal behavior within 2 years prior to study entry
* Pregnant or breastfeeding
* Physiologically dependent on any drugs other than nicotine or marijuana
* History of schizophrenia, bipolar disorder, or other psychotic disorders
* Currently taking cough medicine (e.g., dextromethorphan) and/or albuterol

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2004-06; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Herbert Kleber, MD, Principal Investigator — New York State Psychiatric Institute
Locations (1):
- Research Foundation for Mental Hygiene, Inc., New York, New York, United States

REFERENCES:
- See also: Click here for the Substance Treatment and Research Service website — http://www.stars.columbia.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were seeking treatment for problems related to cocaine use and were recruited by local advertising/referrals in the New York City area. Two types of adS were placed: (1) ads for treatment of cocaine dependence, and (2) ads for treatment for cocaine dependence and possible problems with inattention and/or hyperactivity.
Groups:
- Atomoxetine: Initially, atomoxetine was administered at 20 mg/day for three days. This dose was then increased to 40 mg/day for four days. During the second week of the trial, the dose was increased to 60 mg/day and later increased to 80 mg/day at the start of Week 3. Patients were then maintained at 80 mg per day for four weeks. At the beginning of Week 7, patients were maintained at 80 mg/day or increased to the maximal dose of 100 mg/day if there was less than a 50% reduction of ADHD symptoms (as determined by the Adult ADHD Rating Scale; Murphy, 1996) and if the patients were tolerating the medication well. They were then maintained at 80 mg/day or 100 mg/day for the remaining six weeks of the trial. All patients received two capsules to be taken once a day in the morning.
Period: Overall Study
Arm/Group | Atomoxetine
Started | 20
Completed | 5 (13 reached the maintenance dose phase of treatment; 9 completed at least six weeks of treatment.)
Not Completed | 15
Not completed — Lost to Follow-up | 8
Not completed — relocated | 1
Not completed — Withdrawal by Subject | 1
Not completed — Physician Decision | 3
Not completed — Adverse Event | 2

BASELINE CHARACTERISTICS:
Arm/Group | Atomoxetine
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.3 (6.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 19
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: the Adult ADHD Rating Scale (AARS) (30% Reduction)
Description: AARS is a self report that measures symptoms of adult ADHD. The primary outcome was the percentage of patients achieving a 30% reduction from baseline on the AARS scale. The AARS is scored on a continuous, range 0-54. 0 being no symptoms and 54 being indicative of the most severe level of symptoms.
Time Frame: baseline compared to rating at week 12 or last rating during study participation
Population: All participants
Measure: Number; unit: percent of participants
Arm/Group | Atomoxetine
Number analyzed (Participants) | 20
percent of participants | 50

2. Primary Outcome: ADHD Symptoms Based on Adult ADHD Rating Scale Scale (AARS)
Description: Weekly AARS scores (continuous, range 0-54) were examined with the baseline score compared to that at the last assessment obtained and change in these scores over time. The AARS looks at adult ADHD symptoms. A score of 0 represents no symptoms and 54 would be indicative of the most severe level of symptoms.
Time Frame: measured during 12 weeks or length of study participation
Population: Comparing overall baseline scores to end of study scores for patients who had at least two AARS weekly measures completed
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Atomoxetine
Number analyzed (Participants) | 18
scores on a scale
  baseline | 31.4 (9.8)
  end of study | 21.2 (12.4)

ADVERSE EVENTS:
Time Frame: 12 weeks or length of study participation
Arm/Group | Atomoxetine
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 5/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atomoxetine (N=20)
nausea (Gastrointestinal disorders) | 2 (2)
headache (General disorders) | 1 (1)
chest pain (Cardiac disorders) | 1 (1)
anxiety (Psychiatric disorders) | 2 (2)
dizziness (General disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Clearly, there are limitations of this study including the high drop-out rate, small sample size, and lack of a control group.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes